CLINICAL TRIAL: NCT06957184
Title: A Comparison Between Bladder Dissection Before and After Uterine Incision During Cesarean Section for Placenta Accreta Spectrum: A Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: bladder disection in PAS
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): 40 patients will have bladder dissection at the start of caesarean section for patient with morbidly adherent placenta
  Interventions: Procedure: bladder dissection in placenta accreta spectrum
- group b (Active Comparator): 40 patients will have bladder dissection after closing uterine incision and just before clamping uterine artery in case of caesarean hysterectomy
  Interventions: Procedure: bladder dissection in placenta accreta spectrum

INTERVENTIONS:
Procedure: bladder dissection in placenta accreta spectrum — All caesarean sections will be performed by a surgeon who has experience in performing caesarean hysterectomy in both groups.
  * Scrubbing the abdomen as usual.
  * Subumblical midline skin incision versus Pfannenstiel incision will be chosen according to site of the placenta and previous surgeries.
  * In group A careful bladder dissection will be done before uterine incision with ensuring hemostasis, uterine incision will be done above the placenta, after delivering the baby awaiting for placental separation if not proceeding for caesarean hysterectomy.
  * In group B uterine incision will be done above the placenta and after delivering the baby awaiting for placental separation if not proceeding to caesarean hysterectomy and dissecting bladder just before clamping uterine artery.

SUMMARY:
The worldwide incidence of placenta accreta spectrum is increasing, following the trend of rising caesarean delivery. It is an heterogeneous condition associated with a high maternal morbidity and mortality rate (Jauniaux et al., 2018).

caesarean hysterectomy is considered the gold standard for the treatment of placenta accreta. Also this radical approach is associated with high rates of severe maternal morbidity as hemorrhage and insult to surrounding organs during surgery (Hoffman et al., 2010).

Surgeons should be able to dissect the bladder safely and confidently through minimally invasive techniques, to avoid surgical injury, it is important to use anatomic landmarks, minimize the use of cauterization (Farhat and Casale, 2018).

All centers are encouraged to develop guidelines to manage the potential urologic complications of these cases tailored to their resources (Taneja and Shah, 2017).

This study aims to evaluate the timing of bladder dissection in caesarean section in patient with placenta accreta spectrum.

DETAILED DESCRIPTION:
Objective:

Try to provide preliminary data to judge between two different approaches during caesarean section for morbidly adherent placenta, that's are bladder dissection before and after uterine incision as regard operative time, blood loss, and incidence of urological injuries.

Research Question:

- Does bladder dissection after uterine incision in caesarean sections with PAS avoids bladder injuries compared to bladder dissection before uterine incision and does it affects operative time and blood loss.

Research hypothesis:

* Null Hypothesis (H₀): There is no significant difference in performing bladder dissection prior nor after uterine incision in caesarean sections with PAS
* Alternative Hypothesis (H₁):. bladder dissection before uterine incision in caesarean sections with PAS has superior outcomes compared to bladder dissection after uterine incision.

ELIGIBILITY:
Inclusion Criteria:

* Women with BMI at or under 35kg/m2
* Women with history of at least previous two caesarean section
* Gestational age more than 32 weeks with viable fetus.
* Women with any degree of placenta previa.
* Women with placenta falling in the PAS.
* Willing and able to provide informed consent.

Exclusion Criteria:

* o History of urinary bladder injury.

  * History of urinary or renal disorders
  * Women with coagulation disorders or on anticoagulation therapy.
  * Patients who are hemodynamically unstable before skin incision

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
o Blood loss | 1 year
  assessed by number of soaked towels and suction reservoir)

CONTACTS AND LOCATIONS:
Overall Officials: khaled saed, professor, Study Director — direcror

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eller AG, Porter TF, Soisson P, Silver RM. Optimal management strategies for placenta accreta. BJOG. 2009 Apr;116(5):648-54. doi: 10.1111/j.1471-0528.2008.02037.x. Epub 2009 Feb 4. PMID 19191778
- [Background] Hoffman MS, Karlnoski RA, Mangar D, Whiteman VE, Zweibel BR, Lockhart JL, Camporesi EM. Morbidity associated with nonemergent hysterectomy for placenta accreta. Am J Obstet Gynecol. 2010 Jun;202(6):628.e1-5. doi: 10.1016/j.ajog.2010.03.021. PMID 20510963
- [Background] Jauniaux E, Collins S, Burton GJ. Placenta accreta spectrum: pathophysiology and evidence-based anatomy for prenatal ultrasound imaging. Am J Obstet Gynecol. 2018 Jan;218(1):75-87. doi: 10.1016/j.ajog.2017.05.067. Epub 2017 Jun 24. PMID 28599899
- [Background] Marshall NE, Fu R, Guise JM. Impact of multiple cesarean deliveries on maternal morbidity: a systematic review. Am J Obstet Gynecol. 2011 Sep;205(3):262.e1-8. doi: 10.1016/j.ajog.2011.06.035. Epub 2011 Jun 15. PMID 22071057
- See also: pubmed — http://pubmed.ncbi.nlm.nih.gov/22071057/